CLINICAL TRIAL: NCT00111813
Title: Phase I Clinical Trial of Vorinostat (MK-0683) in Combination With Bortezomib in Patients With Advanced Multiple Myeloma
Brief Title: Phase 1 Study of Vorinostat and Bortezomib in Multiple Myeloma (MK-0683-015 EXT 1 (AM1))
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-015; 2005_018
Record Dates: First submitted 2005-05-25; First posted 2005-05-26 (Estimated); Results first posted 2011-04-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Vorinostat; Bortezomib

ARMS (6):
- vorinostat 200 mg + bortezomib 0.7 mg/m^2 (Experimental): Vorinostat capsules given twice daily (b.i.d.); bortezomib injection given on Days 4, 8, 11, and 15 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib
- vorinostat 200 mg + bortezomib 0.9 mg/m^2 (Experimental): Vorinostat capsules given b.i.d.; bortezomib injection given on Days 4, 8, 11, and 15 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib
- vorinostat 300 mg + bortezomib 1.3 mg/m^2 (Experimental): Vorinostat given once daily (q.d.); bortezomib given on Days 1, 4, 8, and 11 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib
- vorinostat 400 mg + bortezomib 0.9 mg/m^2 (Experimental): Vorinostat given q.d.; bortezomib given on Days 1, 4, 8, and 11 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib
- vorinostat 400 mg + bortezomib 1.1 mg/m^2 (Experimental): Vorinostat given q.d.; bortezomib given on Days 1, 4, 8, and 11 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib
- vorinostat 400 mg + bortezomib 1.3 mg/m^2 (Experimental): Vorinostat given q.d.; bortezomib given on Days 1, 4, 8, and 11 of each cycle.
  Interventions: Drug: vorinostat; Drug: bortezomib

INTERVENTIONS:
Drug: vorinostat — Vorinostat capsules. Treatment in 21 day cycles (participants receive vorinostat for 14 days followed by a 7 day break).
  Other Names: MK0683; Zolinza®; Suberoylanilide Hydroxamic Acid (SAHA)
Drug: bortezomib — Bortezomib injection. Given twice weekly for 2 weeks with a 1 week break. Treatment in 21 day cycles.
  Other Names: Velcade

SUMMARY:
The purposes of this study are:

* To determine the maximum tolerated dose (MTD) for the combination of oral vorinostat and bortezomib in participants with advanced multiple myeloma
* To assess the safety and tolerability of this regimen and to document the participant's clinical status (by anti-tumor activity) for this combination, as determined per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adults with refractory or relapsed multiple myeloma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (a measurement to determine participant's ability to perform daily activities)
* Adequate bone marrow reserve
* Adequate hepatic and renal function
* Ability to swallow capsules
* 3 weeks or more since prior chemotherapy and have recovered from prior toxicities

Exclusion Criteria:

* Participants who plan to have a bone marrow transplant within 4 weeks of start of treatment
* Participants with prior treatment with other investigational agents with a similar anti-tumor mechanism
* Participants with other active/uncontrolled clinically significant illness
* Pregnant or nursing female participants
* Participants who received bortezomib within 3 months of start of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Weber DM, Graef T, Hussein M, Sobecks RM, Schiller GJ, Lupinacci L, Hardwick JS, Jagannath S. Phase I trial of vorinostat combined with bortezomib for the treatment of relapsing and/or refractory multiple myeloma. Clin Lymphoma Myeloma Leuk. 2012 Oct;12(5):319-24. doi: 10.1016/j.clml.2012.07.007. PMID 23040438

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat 200 mg + Bortezomib 0.7 mg/m^2: Vorinostat capsules given twice daily (b.i.d.). Treatment in 21 day cycles (participants received vorinostat for 14 days followed by a 7 day break).
  Bortezomib injection. Treatment in 21 day cycles (participants received bortezomib on Days 4, 8, 11, and 15 of each cycle).
- Vorinostat 200 mg + Bortezomib 0.9 mg/m^2: Vorinostat capsules given b.i.d. Treatment in 21 day cycles (participants received vorinostat for 14 days followed by a 7 day break).
  Bortezomib injection. Treatment in 21 day cycles (participants received bortezomib on Days 4, 8, 11, and 15 of each cycle).
- Vorinostat 300 mg + Bortezomib 1.3 mg/m^2: Vorinostat capsules given once daily (q.d.). Treatment in 21 day cycles (participants received vorinostat for 14 days followed by a 7 day break).
  Bortezomib injection. Treatment in 21 day cycles (participants received bortezomib on Days 1, 4, 8, and 11 of each cycle).
- Vorinostat 400 mg + Bortezomib 0.9 mg/m^2; Vorinostat 400 mg + Bortezomib 1.1 mg/m^2; Vorinostat 400 mg + Bortezomib 1.3 mg/m^2: Vorinostat capsules given q.d. Treatment in 21 day cycles (participants received vorinostat for 14 days followed by a 7 day break).
  Bortezomib injection. Treatment in 21 day cycles (participants received bortezomib on Days 1, 4, 8, and 11 of each cycle).
Period: Overall Study
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Started | 3 | 3 | 10 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 3 | 3 | 10 | 5 | 6 | 6
Not completed — Adverse Event | 1 | 2 | 4 | 2 | 2 | 2
Not completed — Progressive disease | 2 | 1 | 5 | 3 | 4 | 3
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Vorinostat capsules given 200 mg b.i.d., 300 mg q.d., or 400 mg q.d. Treatment in 21 day cycles (participants received vorinostat for 14 days followed by a 7 day break).
  Bortezomib injection. Treatment in 21 day cycles (participants received bortezomib 0.7 mg/m^2, 0.9 mg/m^2, 1.1 mg/m^2, or 1.3 mg/m^2 twice weekly on Days 1, 4, 8, and 11 or on Days 4, 8, 11, and 15 of each cycle, depending on dose level.
Arm/Group | All Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Treatment With Vorinostat
Description: Event causing discontinuation from the study was defined as (1) progressive disease OR (2) intolerable toxicity.
  Progressive disease was defined as:
  * >25% increase in the level of serum monoclonal paraprotein.
  * 25% increase in 24-hour urinary light chain excretion.
  * >25% increase in plasma cells in a bone marrow aspirate or on trephine
  biopsy.
  * Development of new bone lesions or soft tissue plasmacytomas.
  * Development of hypercalcemia.
  Intolerable toxicity was based on the clinical judgment of the investigator.
Time Frame: Day 1 to an event causing discontinuation from the study, assessed up to 29 months
Measure: Mean (Full Range); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 34
Days
  200 mg | 4.6 [1 to 15]
  300 mg | 72.6 [28 to 210]
  400 mg | 107.1 [11 to 496]

2. Secondary Outcome: Number of Participants With Dose Modifications of Either Vorinostat or Bortezomib Due to Adverse Experiences (AEs) After Treatment With Study Drug
Description: An adverse experience (AE) was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the sponsor's product, was also an adverse experience.
Time Frame: Day 1 to disease progression, toxicity, or death, assessed up to 29 months
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10 | 6 | 6 | 6
Participants
  No dose modification | 3 | 3 | 8 | 4 | 3 | 3
  One dose modification | 0 | 0 | 2 | 2 | 1 | 0
  Two or more dose modifications | 0 | 0 | 0 | 0 | 2 | 3

3. Secondary Outcome: Mean Time to First AE Resulting in a Dose Modification in Either Vorinostat or Bortezomib
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the sponsor's product, was also an adverse experience.
Time Frame: Day 1 to disease progression, toxicity, or death, assessed up to 29 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10 | 6 | 6 | 6
Days | NA (NA) — No participants had a dose modification at this dose. | NA (NA) — No participants had a dose modification at this dose. | 58 (39) | 58 (11) | 128 (148) | 32 (5)

4. Secondary Outcome: Clinical AE Summary
Description: An AE was defined as any unfavorable/unintended change in the structure/function/chemistry of the body temporally associated with the use of study drug, or any worsening of a preexisting condition.
  A serious AE (SAE) was any AE that resulted in death, was life threatening, resulted in a persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a new cancer, or was an overdose.
Time Frame: Day 1 up to disease progression, toxicity, or death, assessed up to 30 days after end of treatment (up to 30 months)
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10 | 6 | 6 | 6
Participants
  With one or more AEs | 3 | 3 | 10 | 6 | 6 | 6
  With no AEs | 0 | 0 | 0 | 0 | 0 | 0
  With drug-related AEs | 2 | 3 | 10 | 6 | 6 | 6
  With Serious AEs (SAEs) | 0 | 1 | 2 | 4 | 4 | 2
  With drug-related SAEs | 0 | 0 | 1 | 4 | 2 | 1
  Who died | 0 | 0 | 0 | 0 | 0 | 0
  Who discontinued due to AEs | 1 | 2 | 4 | 2 | 1 | 2
  Who discontinued due to drug-related AEs | 0 | 2 | 3 | 2 | 1 | 1
  Who discontinued due to SAEs | 0 | 0 | 1 | 2 | 0 | 1
  Who discontinued due to drug-related SAEs | 0 | 0 | 1 | 2 | 0 | 0

5. Secondary Outcome: Laboratory AE Summary
Description: An AE was defined as any unfavorable/unintended change in the structure/function/chemistry of the body temporally associated with the use of study drug, or any worsening of a preexisting condition.
  A SAE was any AE that resulted in death, was life threatening, resulted in a persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a new cancer, or was an overdose.
  A lab (S)AE was any lab value considered clinically significant in the investigator's judgment.
Time Frame: Day 1 up to disease progression, toxicity, or death, assessed up to 29 months
Measure: Number; unit: Participants
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Number analyzed (Participants) | 3 | 3 | 10 | 6 | 6 | 6
Participants
  With one or more laboratory AEs | 1 | 1 | 3 | 0 | 2 | 3
  With no laboratory AEs | 2 | 2 | 7 | 6 | 4 | 3
  With drug-related laboratory AEs | 1 | 0 | 2 | 0 | 1 | 3
  With laboratory Serious AEs (SAEs) | 0 | 0 | 0 | 0 | 0 | 0
  With drug-related laboratory SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Who died | 0 | 0 | 0 | 0 | 0 | 0
  Who discontinued due to laboratory AEs | 0 | 0 | 0 | 0 | 0 | 0
  Who discontinued due to drug-related lab AEs | 0 | 0 | 0 | 0 | 0 | 0
  Who discontinued due to laboratory SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Who discontinued due to drug-related lab SAEs | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/10 | 4/6 | 4/6 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 10/10 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 (N=3) | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 (N=3) | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 (N=10) | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 (N=6) | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 (N=6) | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2 (N=6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat 200 mg + Bortezomib 0.7 mg/m^2 (N=3) | Vorinostat 200 mg + Bortezomib 0.9 mg/m^2 (N=3) | Vorinostat 300 mg + Bortezomib 1.3 mg/m^2 (N=10) | Vorinostat 400 mg + Bortezomib 0.9 mg/m^2 (N=6) | Vorinostat 400 mg + Bortezomib 1.1 mg/m^2 (N=6) | Vorinostat 400 mg + Bortezomib 1.3 mg/m^2 (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 5 (12) | 2 (3) | 5 (19) | 4 (7)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (15) | 2 (3) | 2 (4)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Scintillating scotoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (7) | 3 (11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (5) | 8 (13) | 4 (18) | 6 (36) | 6 (17)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (12) | 6 (13) | 5 (24) | 3 (19) | 6 (24)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (7) | 3 (7) | 3 (4) | 5 (8)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 3 (6) | 5 (12) | 6 (20) | 2 (11) | 5 (33)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Metaplasia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (5)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 2 (2) | 2 (2)
Ulcer (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (6) | 2 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 0 (0) | 2 (4)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypouricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3) | 2 (2)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (3) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (6) | 1 (7) | 2 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (8) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (3) | 1 (1) | 3 (6) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (2) | 5 (8) | 2 (3) | 1 (2) | 1 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 2 (5) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (5)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as

confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.